CLINICAL TRIAL: NCT00649181
Title: Single-Dose Fasting In Vivo Bioequivalence Study of Metolazone Tablets (5 mg; Mylan) and Zaroloxyn® Tablets (5 mg; Celltech) in Healthy Volunteers
Brief Title: Fasting Study of Metolazone Tablets 5 mg and Zaroloxyn® Tablets 5 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: METO-0361
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Metolazone

ARMS (2):
- 1 (Experimental): Metolazone Tablets 5 mg
  Interventions: Drug: Metolazone Tablets 5 mg
- 2 (Active Comparator): Zaroloxyn® Tablets 5 mg
  Interventions: Drug: Zaroloxyn® Tablets 5 mg

INTERVENTIONS:
Drug: Metolazone Tablets 5 mg — 2x5mg, single dose fasting
  Arms: 1
Drug: Zaroloxyn® Tablets 5 mg — 2x5mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan metolazone 5 mg tablets to Celltech Zaroxolyn® 5 mg tablets following a single, oral 10 mg (2 x 5 mg) dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older
2. Sex: Male and/or non-pregnant, non-lactating female

   1. Women of childbearing potential must have negative serum -human chorionic gonadotropin (β-HCG) pregnancy tests performed within 14 days prior to the start of the study and on the evening prior to each dose administration. If dosing is scheduled on Sunday or Monday, serum samples for β-HCG testing may be collected and sent for analysis within 48 hours prior to dosing for both study periods. An additional serum (Beta-HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or use an acceptable form of contraception throughout the duration of the study. No hormonal contraceptives or hormonal replacement therapy are permitted in this study. Acceptable forms of contraception include the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. surgical sterility (tubal ligation, oophorectomy or hysterectomy) or postmenopausal accompanied with a documented postmenopausal course of at least one year.
   3. During the course of the study, from study screen until study exit - including the washout period, women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive device. This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs.) for men and 48 kg (106 lbs.) for women and within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, 12-lead ECG, Hepatitis B, Hepatitis C and HIV tests, and urine drug screen including amphetamine, benzodiazepine, cannabinoid, cocaine, opiate screen, and phencyclidine) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within one year prior to dosing.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
3. Medications:

   1. Use of any medication within the last 14 days prior to the initial dose of study medication, including over-the-counter medications.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
   3. Use of hormonal contraceptives and hormonal replacement therapy within three months prior to the initial dose of study medication.
4. Diseases:

   a. History of any significant chronic disease and/or hepatitis. b. History of drug and/or alcohol abuse. d. Acute illness at the time of either the pre-study medical evaluation or dosing.

   e. A positive HIV, Hepatitis B, or Hepatitis C test result.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to metolazone, sulfonamide-derived drugs, thiazides, quinethazone or other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Clark, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html